CLINICAL TRIAL: NCT05819411
Title: Stigma-Treatment Enhanced Incentivized Directly Observed Therapy for People With HIV Who Inject Drugs
Brief Title: Intervention to Improve HIV Self-care Among People Who Inject Drugs
Acronym: iSTRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Fenway Community Health (Other); National Institute on Drug Abuse (NIDA) (NIH); Boston University (Other)
Responsible Party: Principal Investigator, Abigail Batchelder, Ph.D., M.P.H., Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002094; R34DA053686 (NIH)
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Hiv; Substance Use Disorders
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This intervention includes 6 face-to-face therapy sessions with a trained clinician plus an incentivized directly observed therapy (iDOT) intervention facilitated via a mobile application.
  Interventions: Behavioral: Project iSTRIVE; Behavioral: incentivized Directly Observed Therapy (iDOT)
- incentivized Directly Observed Therapy (iDOT) (Active Comparator): Participants in the iDOT condition will be provided a mobile application to facilitate video recording of their daily medication adherence in order to receive small, escalating monetary incentives for HIV medication adherence.
  Interventions: Behavioral: incentivized Directly Observed Therapy (iDOT)

INTERVENTIONS:
Behavioral: Project iSTRIVE — This intervention includes 6 face-to-face therapy sessions with a trained clinician to develop skills to counter internalized stigma and shame as barriers to HIV self-care. Both the intervention group and the active control group will also receive a mobile app-based iDOT intervention.
  Arms: Intervention
Behavioral: incentivized Directly Observed Therapy (iDOT) — Both the intervention group and the active control group will receive a mobile app-based iDOT intervention.

SUMMARY:
This study will implement a pilot randomized controlled trial (RCT, N=50) to refine and assess the feasibility and acceptability of an emotion regulation and communication skills intervention designed to improve engagement in HIV-care among HIV+ people who report opioid and/or stimulant use and are sub-optimally engaged in HIV care.

DETAILED DESCRIPTION:
Eligible study participants will be screened and enrolled at Fenway Health (Boston, MA). All participants will receive substance use treatment referral information if interested. Participants will be randomized to one of two treatment arms. Participants in both arms will receive a mobile application-facilitated incentivized directly observed therapy (iDOT) intervention. Participants in the control arm will receive iDOT alone. Participants in the intervention arm will receive iDOT in combination with the iSTRIVE intervention. After randomization, participants in the iSTRIVE intervention group will be offered 6 therapy sessions focused on behavioral strategies for improving HIV self-care, meta-cognitive awareness of emotions and thoughts, cognitive restructuring, and assertive communication skills. Participants in the iSTRIVE intervention arm will also receive messages containing customized compassionate self-statements to enhance HIV-related self-care. All participants will be compensated for every research visit and adherence to the iDOT protocol.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* HIV virally unsuppressed (>20 copies/mL) in past year or no past-year HIV viral load result
* Opioid and/or stimulant use behavior endorsed in past 6 months
* Able to provide informed consent
* 18 years or older
* English speaking

Exclusion Criteria:

* HIV negative
* Denying drug use in past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of iSTRIVE intervention | change from baseline to 12 weeks after intervention completion
  Percent of sessions completed (≥70% considered indicative of feasibility).
Feasibility of iDOT intervention | change from baseline to 12 weeks after intervention completion
  Percent of DOT video check ins completed by participants (≥50% considered indicative of feasibility).
Acceptability of intervention | 12 weeks after intervention completion
  A qualitative analysis of exit interviews conducted with iSTRIVE study intervention participants.

SECONDARY OUTCOMES:
HIV Viral Load | change from baseline to 12 weeks after intervention completion
  Viral suppression (≤20 copies/mL) will be assessed via blood draw at the final follow up visit and will be the primary outcome variable in the planned subsequent efficacy trial.
Substance Use | change from baseline to 12 weeks after intervention completion
  Addiction Severity Index-Lite will be used to assess self-reported substance use at each research visit and a subset of questions will be asked at all intervention visits. The primary metric will be number of days a participant reports experiencing drug problems in the past month (0-30), with a decrease in days (i.e., lower number) indicating a favorable outcome.
Injection Drug Use Behaviors | change from baseline to 12 weeks after intervention completion
  We will assess injection behaviors associated with HIV risk by self-report by adapting items identified by Shahesmaeili et al. (Brief Scale to Measure HIV Transmission Risk Among Injecting Drug Users). These questions will include injection behaviors and related factors that differ by gender (e.g., needle borrowing, ancillary equipment sharing, being injected by someone else, and whether injection partners are also sexual partners). The total scale is scored from 0-36, with lower scores indicating favorable outcomes (i.e., reduction in HIV risk behavior).

CONTACTS AND LOCATIONS:
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No